CLINICAL TRIAL: NCT01139892
Title: Canadian Study on the Endovascular Treatment of Unruptured Intracranial Aneurysms Versus Surgical Treatment. A Randomized Comparison of Clinical and Angiographic Results of Intracranial Aneurysms
Brief Title: The Canadian UnRuptured Endovascular Versus Surgery Trial (CURES)
Acronym: CURES
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: ND09.282; CIHR; MOP119554 (Other Grant/Funding Number: Grant to CHUM Research Centre to Dr. Jean Raymond.)
Record Dates: First submitted 2010-06-02; First posted 2010-06-09 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Intracranial Aneurysms
Keywords: Unruptured aneurysm; endovascular treatment; surgical treatment; randomized; intracranial aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgical management: Surgical clipping will be performed within 6 weeks of randomization, according to standards of practice, and under general anaesthesia. Aneurysms thought by the treating physicians to require deliberate permanent proximal vessel occlusion, bypasses, and other flow-redirecting treatments that do not directly clip the aneurysm will not be included.
  Interventions: Procedure: Surgical management
- Endovascular management: Endovascular treatment will be performed within 6 weeks of randomization, according to standards of practice, and under general anaesthesia. Details regarding type of coils, use of adjunctive techniques such as balloon-remodeling or stents, as well as post-treatment medical management issues, will be left up to the physician performing the endovascular treatment.
  Interventions: Procedure: Endovascular management

INTERVENTIONS:
Procedure: Surgical management
  Other Names: Arm 1: clipping
  Groups: Surgical management
Procedure: Endovascular management
  Other Names: Arm 2: coiling
  Groups: Endovascular management

SUMMARY:
Purpose:

Phase 1: (Pilot Phase)

To compare the treatment efficacy of surgical clipping and endovascular coiling for unruptured intracranial aneurysms.

To obtain better estimates of morbidity and mortality related to a surgical or endovascular treatment strategy at one year within the context of an RCT.

To show that an RCT comparing the morbidity and mortality of a surgical management strategy to an endovascular management strategy is feasible.

Phase 2:

To compare the results of surgical and endovascular management strategies, in terms of:

1. Overall mortality and morbidity at 1 and 5 years.
2. The clinical efficacy and safety of a surgical or endovascular management strategy at 1 and 5 years

Hypotheses: Phase 1 Hypotheses:

1. Surgical clipping of intradural, saccular, unruptured intracranial aneurysms is superior to endovascular management in terms of a lesser number of patients experiencing treatment failure.
2. An RCT comparing the clinical outcomes of a surgical versus endovascular management strategy is feasible.

Phase 1 Primary End-points:

• Treatment failure, hereby defined as having occurred when either: the intended initial modality (surgical or endovascular) fails to occlude the aneurysm, a "major" (saccular) angiographic aneurysm recurrence is found, or an intracranial hemorrhagic event occurs during the 1-year follow-up period.

Phase 1 Secondary End-points:

1. Overall morbidity and mortality at one year.
2. Occurrence of morbidity (mRS >2) or mortality following treatment.
3. Occurrence of failure of aneurysm occlusion using the initial intended treatment modality.
4. Occurrence of a "major" (saccular) angiographic aneurysm recurrence.
5. Occurrence of an intracranial hemorrhage following treatment.
6. Peri-treatment hospitalization lasting more than 5 days
7. Discharge following treatment to a location other than home

Treatment:

Trial feasibility, or the capacity for patient recruitment, would require enrollment of at least 8 patients per actively recruiting center per year.

Phase 2 Hypotheses:

It may be too early to explicitly define the primary hypothesis of Phase 2, however, the intent of Phase 2 can be expressed as:

1. One management strategy is superior to the other in terms of clinical outcome at five years.
2. One management strategy is superior to the other in terms of clinical efficacy at five years.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with at least 10 years of remaining life expectancy
* At least one documented, intradural, saccular intracranial aneurysm
* The patient and aneurysm are considered appropriate for either surgical or endovascular treatment by the treating team
* Aneurysm size 3-25 mm

Exclusion Criteria:

* Patients with any intracranial hemorrhage, including SAH, within the previous 30 days
* Lesion characteristics not readily suitable for either endovascular or surgical treatment, in the opinion of the physician(s) intending to treat the aneurysm
* Multiple aneurysms, where the treatment plan includes both surgical clipping as well as endovascular coiling
* Aneurysm anticipated (pre-operatively) to require proximal vessel occlusion, a bypass, or other flow-redirecting therapy (such as flow-diverting stents) as part of treatment plan
* Patients with baseline mRS >2
* Patients with a single cavernous aneurysm
* Patients with dissecting, fusiform, or mycotic aneurysms
* Patients with AVM-associated aneurysms
* Pregnant patients (randomization (and treatment) may be delayed until after delivery)
* Patients with absolute contraindications to anaesthesia, endovascular treatment or administration of contrast material, including low-osmolarity agents or gadolinium
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2010-09-26 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Treatment failure | One Year
  Defined as having occurred when either: the intended initial modality (surgical or endovascular) fails to occlude the aneurysm, a "major" (saccular) angiographic aneurysm recurrence is found, or an intracranial hemorrhagic event occurs during the 1-year follow-up period.

SECONDARY OUTCOMES:
Morbidity and mortality: 2. Hospitalization >5 days : physician reporting. 3. Discharge other than to home: physician reporting. | one year
  Overall morbidity and mortality at one year. Morbidity = modified Rankin scale score >2. The Modified Rankin Scale score will be determined by an independent health-care professional, not directly involved in the CURES study, and blinded to treatment allocation.
Occurrence of morbidity (mRS >2) or mortality following treatment. | 6 weeks post-treatment
  Occurrence of morbidity (mRS >2) or mortality following treatment. The Modified Rankin Scale score will be determined by an independent health-care professional, not directly involved in the CURES study, and blinded to treatment allocation.
Failure of aneurysm occlusion | 1 year
  Occurrence of failure of aneurysm occlusion using the initial intended treatment modality as determined by the local treating physician. Patients left with clinically concerning aneurysm residuals (in the opinion of the treating physician) after the treatment attempt will count as a failure of the initial treatment.
  In the surgically-treated patients, the surgeon's judgment of whether or not the aneurysm is fully occluded with the clip will be used to determine failure of aneurysm occlusion. Because the primary end-points in Phase 1 is a composite end-point, it does not distinguish between aneurysm remnants found immediately post-treatment (failure to completely occlude the aneurysm) and recurrences (or residuals) found at one-year post-treatment. Even if a surgically-treated aneurysm felt to be completely occluded by the surgeon is in fact inadequately treated, this will be found at the one year follow-up imaging mark, and thus does not constitute a source of bias.
Occurrence of a "major" (saccular) angiographic aneurysm recurrence. | 1 year
  Occurrence of a "major" (saccular) angiographic aneurysm recurrence.
Occurrence of an intracranial hemorrhage | 1 year
  Determined using non-invasive angiography (CTA or MRA) performed at 12 +/- 2 months post-treatment, with all images sent to CURES headquarters for Core Lab confirmation. This follow-up imaging is considered to be part of normal follow-up after aneurysm treatment. Although CTA and MRA are known to have different sensitivities in detecting aneurysm remnants, both modalities are equally well-suited to the discovery of what we are looking for: a concerning, saccular aneurysm residual or remnant. Because the definition of "major", "concerning", or "saccular" aneurysm residual or remnant remains subjective, (as does the threshold for re-treatment) local investigators will be requested to record the occurrence of what they consider to be a "major" saccular recurrence, but the final determination of this end-point will be determined by an independent Core Lab.
Hospitalization lasting more than 5 days | 6-weeks post-treatment
  This end-point will be recorded by the local treating physician on discharge.
Discharge following treatment to a location other than home | 6-weeks post-treatment
  This end-point will be recorded by the local treating physician on discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Darsaut, MD, Principal Investigator — University of Alberta; Jean Raymond, MD, Principal Investigator — Université de Montréal
Locations (6):
- Centre hospitalier universitaire de Liège, Liège, Belgium
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - Centre hospitalier de l'Université de Montréal - CHUM, Montreal, Quebec
- CHRU de Lille, Lille, France

REFERENCES:
- [Derived] Naggara O, Darsaut T, Trystram D, Tselikas L, Raymond J. Unruptured intracranial aneurysms: why we must not perpetuate the impasse for another 25 years. Lancet Neurol. 2014 Jun;13(6):537-8. doi: 10.1016/S1474-4422(14)70091-2. No abstract available. PMID 24849854